CLINICAL TRIAL: NCT03603509
Title: Transcriptomic Signatures of Influenza Vaccine Responses
Brief Title: Gene Signatures of Influenza Vaccine Responses in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Richard B. Kennedy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-010601; R01AI132348 (NIH)
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Influenza
Keywords: Fluad, MF59, Fluzone, HDFlu, Influenza, Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine; Fluzone High-Dose; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Eligible subjects who consent and enroll will be randomly assigned to receive either the Fluad Vaccine or Fluzone High-Dose vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluad vaccine (Active Comparator): Subjects receive a single dose of the Fluad influenza vaccine.
  Interventions: Drug: Fluad Vaccine
- Fluzone vaccine (Active Comparator): Subjects receive a single dose of the Fluzone High-Dose influenza vaccine.
  Interventions: Drug: Fluzone High-Dose

INTERVENTIONS:
Drug: Fluad Vaccine — FLUAD is an inactivated influenza vaccine indicated for active immunization against influenza. disease caused by influenza virus subtypes A and type B contained in the vaccine. FLUAD is. approved for use in persons 65 years of age and older.
  Other Names: adjuvanted influenza vaccine
  Arms: Fluad vaccine
Drug: Fluzone High-Dose — FLUZONE® HIGH-DOSE vaccine is indicated for people 65 years of age and older to help prevent influenza disease caused by influenza A and B strains contained in the vaccine.
  Other Names: high dose influenza vaccine
  Arms: Fluzone vaccine

SUMMARY:
The purpose of this research study is to better understand the immune response to the Adjuvanted Subunit flu vaccine (MF59) and the High Dose flu vaccine (HDFlu) in people 65 years of age and older. The research team will be studying why immune response diminishes as people get older in both men and women. The ultimate goal is to understand how flu immunity develops after vaccination. This information may lead to the development of more effective flu vaccines in the future.

DETAILED DESCRIPTION:
The overall goal of this proposal is to determine how vaccine type, sex, and gene expression influence both innate and T helper cell immune responses using systems biology and bioinformatics as tools to comprehensively assess the human transcriptome. We will evaluate sex-dependent immune responses to two unique influenza vaccines in a population of older adults; the recently FDA-licensed MF59-adjuvanted influenza subunit vaccine and the high-dose split virion influenza virus vaccine. The influence of sex on immune response to vaccination has been observed across multiple vaccines (including standard dose influenza vaccines, but the mechanisms are unknown, it affects all age groups regardless of hormonal status, and existing studies focus almost exclusively on humoral immune responses. Relatively little is known about the effect of sex on innate and T helper responses following vaccination and we are unaware of any studies evaluating the effect of sex on immune responses to adjuvanted influenza vaccine. The presence of adjuvant (MF59Flu) or higher antigen (Ag) dose leads to greater immunogenicity through mechanisms that have not been fully deciphered and are likely to be different. Further, a direct comparison of innate and T helper immune responses between adjuvanted and high dose influenza vaccines has not been reported.

The study design will include 200 generally healthy individuals (ages ≥65) who meet all inclusion criteria. 100 subjects will receive each vaccine with equal sex representation in each subgroup (a factorial design for sex by vaccine type). Subjects will undergo venipuncture for blood samples (~100 mL each, sufficient for the proposed assays) before vaccination and at three timepoints after vaccination (Day 1, Day 8, Day 28).

The clinical characterization of our study subjects will include demographic information, height, weight, BMI, waist circumference, medications, and medical conditions that do not meet exclusion criteria (see Protection of Human Subjects). We will also quantify blood leukocyte populations (CBC, WBC differential).

Immunosenescence and cytomegalovirus (CMV) infection can affect influenza vaccine-induced immune responses. We will evaluate whether CMV seropositivity or other measures of immunosenescence are associated with immune response and whether they interact with vaccine type/sex.

We will monitor/characterize transcriptional changes (mRNA and miRNA) as well as measures of immune function (cytokine secretion, leukocyte surface phenotype, hemagglutination inhibiting antibody titer, and memory B cell ELISPOT) at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ages 18-40 or of 65 and or older at the time of enrollment
* Eligible to receive Fluad® (MF59Flu) or Fluzone® (HDFlu) if age 65 or older
* No history of anaphylactic reaction to gelatin, neomycin, or other vaccine component
* Not pregnant
* No immunosuppression or immunodeficiency
* No acute illness at time of vaccination
* Determined by medical history and clinical judgment to be eligible for the study, by being generally healthy, with no autoimmune or immunosuppressive conditions and having stable current medical conditions (subjects with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease 12 weeks before receipt of study vaccine, will be eligible. A change in dose or therapy within a category (e.g., change from one nonsteroidal anti-inflammatory drug to another) is allowed. A change to a new therapy category (e.g., surgery or addition of a new pharmacological class) is only allowed if it is not caused by worsening disease. A change to a new therapy category caused by worsening disease is considered significant and therefore ineligible for enrollment.
* Patients with diabetes mellitus are eligible for inclusion if they have had a hemoglobin A1c measurement of <8.0 within the past 6 months prior to enrollment. These hemoglobin A1c measurements are recommended at least twice yearly by the American Diabetes Association (ADA), and the target levels here are representative of the goals of the ADA. These hemoglobin A1c levels will ensure that these participants have good glycemic control. (American Diabetes Association. American Diabetes Association Position Statement: Standards of Medical Care in Diabetes- 2015. Diabetes Care 2015;38(Suppl. 1): S1-S94)
* Able to follow study procedures in the opinion of the investigator
* Expected to be available for the duration of the study
* Weighs >110 lbs

Exclusion Criteria:

* Known or suspected immunodeficiency or receiving treatment with immunosuppressive therapy including cytotoxic agents or systemic corticosteroids (e.g., for cancer, HIV, or autoimmune disease). If systemic corticosteroids have been administered short term for treatment of an acute illness, subjects will be included if corticosteroid therapy (inhaled, intranasal, and intra-articular corticosteroid therapy is permitted) has been discontinued for at least 30 days.
* Serious chronic medical conditions including metastatic malignancy, severe chronic obstructive pulmonary disease requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, precludes the subject from participating in the study. Diabetic patients will be excluded if they do not have a hemoglobin A1c measurement within the past 6 months or if they had a hemoglobin A1c measurement of an A1c >8.0
* Receipt of any blood products, including immunoglobulin, within 6 months of study enrollment.
* Current anticoagulant therapy or a history of bleeding diathesis that would contraindicate intramuscular (IM) injection. (Note: antiplatelet drugs such as aspirin and clopidogrel are permitted.)
* Receipt of any vaccines within the past 30 days prior to enrollment
* Receipt of the current seasonal influenza vaccine other than in this study
* Acute illness within the last 30 days
* Blood donation within the last 58 days prior to study enrollment
* Any medical condition that would, in the opinion of the investigator, interfere with the evaluation of the study objectives
* Pregnant patients will be excluded
* Any condition (e.g. allergic reaction, Guillain-Barre Syndrome) that precludes their receipt of the influenza vaccine

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kennedy, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Started | 120 | 121
Completed | 117 | 117
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluad Vaccine | Fluzone Vaccine | Total
Number analyzed (Participants) | 120 | 121 | 241
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71.7 [68.2 to 76.2] | 71.4 [67.7 to 75.8] | 71.5 [67.9 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 74 | 152
  Male | 42 | 47 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 118 | 119 | 237
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 119 | 121 | 240
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 120 | 121 | 241

OUTCOME MEASURES:

1. Primary Outcome: Innate Cell IFNa2a Production
Description: Cytokine secretion (interferon alpha 2a) after in vitro stimulation with influenza virus
Time Frame: Baseline, Day 1
Population: The number of samples analyzed is less than the study cohort total because some of the serum samples failed in the assay. These failures were either: results did not meet QC, sample degraded and failed to function in the assay properly.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 106 | 112
pg/mL
  Day 0 Stimulated | 112.3650 [67.6193 to 181.9535] | 131.4214 [87.0718 to 187.8301]
  Day 1 Stimulated | 107.5846 [67.6607 to 189.9629] | 134.9071 [90.1967 to 196.628]

2. Primary Outcome: Hemagglutination Inhibition Ab Titer
Description: Reciprocal of the serum dilution exhibiting no hemagglutination (the larger the number, the more agglutinating antibodies the subject has. A titer of equal to more than 1:40 and above is considered a protective antibody titer)
Time Frame: Baseline and Day 28
Population: The number of samples analyzed is less than the study cohort total because some of the serum samples failed in the HAI assay. These failures were either: results did not meet QC, sample degraded and failed to function in the assay properly.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 117 | 117
Titer
  Day 0: number analyzed (Participants) | 111 | 113
  Day 0 | 40 [20 to 60] | 40 [20 to 80]
  Day 8: number analyzed (Participants) | 111 | 115
  Day 8 | 40 [40 to 80] | 80 [40 to 160]
  Day 28: number analyzed (Participants) | 114 | 116
  Day 28 | 80 [40 to 160] | 80 [40 to 160]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Null Hypothesis: HAI Day 28 - HAI Day 0 for Fluad = HAI Day 28 - HAI Day 0 for Fluzone Alternative Hypothesis: HAI Day 28 - HAI Day 0 for Fluad NE HAI Day 28 - HAI Day 0 for Fluzone; Test type: Superiority; p = 0.062, Wilcoxon (Mann-Whitney)

3. Primary Outcome: T Cell Gene Expression
Description: Gene expression counts. The number shown is the total number of RNA molecules whose sequence matches a human gene. This is a measure of how much gene expression is occurring in the cells in each subject's blood sample.
Time Frame: Baseline, Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Total gene counts
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 109 | 110
Total gene counts
  Day 0 | 36019037 [32656120 to 39665767] | 36566557 [33316917.25 to 39356142.75]
  Day 28 | 34319023 [31763324 to 38266331] | 35360483 [33032560.5 to 39424114.25]

4. Primary Outcome: T Cell miRNA Expression
Description: Next generation sequencing of purified T cells' miRNA
Time Frame: Baseline, Day 8, Day 28
Population: Data was not collected or analyzed
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Innate IFNAR1 Cell Gene Expression
Description: IFNAR1 gene counts (the number of molecules of RNA whose sequence matches the interferon alpha receptor 1 gene that were present in the subject's blood sample).
Time Frame: Baseline, Day 8
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Gene counts
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 109 | 110
Gene counts
  Baseline | 1516 [1263 to 1748] | 1572.5 [1275.5 to 1845.75]
  Day 8 | 1450 [1201 to 1751] | 1562 [1327.25 to 1815.75]

6. Primary Outcome: Innate Cell miRNA Expression
Description: Next generation sequencing of purified innate cells' miRNA
Time Frame: Baseline, Day 1, Day 8
Population: Data was not collected or analyzed
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Memory B Cell ELISPOT
Description: Number of influenza-specific Ab producing memory B cells. Spot Forming Units (SFUs) are the frequency of Ab secreting B cells in an ELISPOT assay.
Time Frame: Day 28
Population: A subset of the total participants' samples were tested to determine the scientific value of this outcome. Based on pre-specified optimization analyses the assay results were highly variable and would not be informative, therefore the assay was not run on all participant samples. Results are reported for the participants' samples that were tested for optimization analyses.
Measure: Median (Inter-Quartile Range); unit: SFUs per 200,000 cells
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 6 | 6
SFUs per 200,000 cells | 5.7 [0.9 to 10.4] | 16.3 [6.8 to 19.2]

8. Secondary Outcome: T Cell ELISPOT Response
Description: influenza-specific, IFNg producing, memory T cells. Spot Forming Units (SFUs) are the frequency of IFN-g secreting T cells in an ELISPOT assay.
Time Frame: Day 28
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: SFUs per 200,000 cells
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 4 | 4
SFUs per 200,000 cells | 14.4 [10.6 to 24.1] | 17.4 [14.4 to 20.4]

9. Secondary Outcome: T Cell Phenotype
Description: Flow cytometry analysis of T cells. The results show the percentage of specific white blood cell types are present in each subject's blood sample. Reported as a % of the total peripheral blood mononuclear cells.
Time Frame: Day 28
Population: A subset of the total participants' samples were tested to determine the scientific value of this outcome. Based on pre-specified optimization analyses, it was determined that results did not capture vaccination-specific responses and would not be useful for the clinical trial, therefore the assay was not run on all participant samples. Results are reported for the participants' samples that were tested for optimization analyses.
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 5 | 4
Percentage
  CD3+ T cells | 44.31 [39.88 to 47.76] | 42.5 [38.22 to 46.22]
  CD4+ T cells | 18.41 [17.49 to 20.49] | 17.98 [15.55 to 21.71]
  CD8+ T cells | 8.73 [6.02 to 9.92] | 10.28 [7.55 to 12.03]

10. Secondary Outcome: Innate Cell Phenotype
Description: Flow cytometry analysis of innate cells. The results show the percentage of classical monocytes in each subject's blood sample. The data are reported as a percentage of the peripheral blood mononuclear cells.
Time Frame: Day 1 (stim)
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 3 | 3
Percentage | 70.1 [69.35 to 73.35] | 93.1 [83.35 to 96.15]

11. Secondary Outcome: CMV Serostatus
Description: Serum CMV-specific IgG level. Number reported as Sample Index (the optical density in an ELISA). The Sample Index is a semi-quantitative measure of how much CMV-specific IgG antibodies are in each subject's blood sample. The values range from 0 to 4. Values between 0 and 3 are relative measures of the amount of antibody (0 = no antibody, 1 = a low level of antibody, 3 = a high level of antibody). Values from 3-4 all reflect high levels of antibody but typically exceed the linear range of the assay and cannot be used to quantify exact amounts of antibody.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Sample Index
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 117 | 117
Sample Index | 2.018 [0.129 to 3.784] | 2.709 [0.181 to 3.858]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Test type: Superiority — null hypothesis: CMV Fluad sample index = CMV Fluzone sample index at Baseline alternate hypothesis: CMV Fluad sample index not equal to CMV Fluzone sample index at Baseline; p = 0.29, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: CD4/CD8 Ratio
Description: Flow cytometry analysis of T cells. The results show the ratio of CD4+ T cells compared to CD8+ T cells present in each subject's PBMCs.
Time Frame: Day 28
Population: This outcome requires data from outcome #9. As outcome #9 was determined to be non-informative and was not run on the entire cohort, we do not have the necessary data to calculate this outcome on the entire cohort. Results are reported for the participants' samples for whom outcome #9 was reported from the optimization analyses.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 5 | 4
Ratio | 2.92 [1.86 to 3.4] | 1.69 [1.34 to 3.46]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 28 days on all participants.
Arm/Group | Fluad Vaccine | Fluzone Vaccine
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/121
Other Adverse Events (participants affected / at risk) | 31/120 | 22/121
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluad Vaccine (N=120) | Fluzone Vaccine (N=121)
Sore Arm (Musculoskeletal and connective tissue disorders) | 16 (16) | 11 (11)
Dizzy (General disorders) | 1 (1) | 2 (2)
Body Aches (Nervous system disorders) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 7 (7) | 2 (2)
Trouble with blood draw (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Cold Symptoms (General disorders) | 5 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Swollen neck gland (General disorders) | 0 (0) | 1 (1)
Allergies (General disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Foot Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bruised Arm (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upset Stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bell's Palsy (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diagnosis of Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Kidney Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elevated Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03603509/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03603509/SAP_003.pdf